CLINICAL TRIAL: NCT02204319
Title: Cold Laser: A Modality to Promote Vulvar Healing and Pain Relief
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: ProHealth Care, Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13-21
Record Dates: First submitted 2014-03-24; First posted 2014-07-30 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-04

CONDITIONS: Vulvar Vestibulitis; Vestibulodynia
Keywords: provoked or non-provoked vulvar vestibulitis; low level laser light device
MeSH Terms: conditions — Vulvar Vestibulitis; Vulvodynia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cold Laser Treatment (Experimental): Cold laser used off of the body over the vulvar involved area. The device to be used in this study is the Erchonia Corporation variable frequency pulsed wave low level laser device employing three independent 7 milliWatt, 635 nanometer red light diodes mounted in a hand-held device and is a variable frequency pulsed wave device. Weekly visits x 6 with 5 minute treatments over vulva and sacral nerve roots each.
  Interventions: Device: Cold laser

INTERVENTIONS:
Device: Cold laser — Erchonia Corporation variable frequency pulsed wave low level laser device employing three independent 7 milliWatt, 635 nanometer red light diodes mounted in a hand-held device and is a variable frequency pulsed wave device.
  Other Names: The Erchonia Laser device

SUMMARY:
The objectives of this pilot study are to demonstrate effectiveness of application of the Erchonia Laser (manufactured by Erchonia Corporation),a non-invasive, non-significant risk low level laser red diode light therapy device, in providing relief of pain symptoms in patients with provoked and non- provoked vulvar vestibulitis; to reduce the frequency of use of oral medications to manage pain symptoms; and to reduce the debilitating affect vulvar vestibulitis has on the patient's daily activities, relationships and emotional well-being.

DETAILED DESCRIPTION:
In the current proposed pilot study, application of a low level laser light device, manufactured by Erchonia Corporation, to reduce the pain of vulvar vestibulitis will be evaluated. The Erchonia Laser device will emit three independent 7 milliWatt, 635 nanometer red light diodes in a hand-held device and is a variable frequency pulsed wave device.

Erchonia low level lasers have been determined safe and effective and non-significant risk (NSR) by the Food and Drug Administration (FDA) for application for numerous and various pain reduction indications, providing justification for the anticipated safety and effectiveness of application of the Erchonia Laser to reduce pain in patients with vulvar vestibulitis. The FDA has granted 510(k) clearances for Erchonia low level laser devices for five pain reduction indications, all cleared under Product Code 'NHN', defined as: "A light based non-laser device that emits energy in infrared or other wavelengths, provides non-heating and non-thermal effect, and is indicated for adjunctive use in pain therapy or related indication. It does not provide therapeutic topical heating."

The research will be conducted at ProHealth Care; Inc. across four campuses. Patients will be seen in private rooms in the therapy departments.

All study staff are licensed in the field of either Occupational Therapy or Physical therapy (2 in each) with the advanced continuing education necessary to call them a "specialist" in the treatment of pelvic floor disorders. All investigators will complete CITI training for research.

Subjects will be referred into the ProHealth Care system via a prescription for pelvic floor therapy signed by a licensed medical professional with the expertise to diagnose Vulvar vestibulitis. Written information regarding the study and proposed treatment will also be mailed to a larger group of pelvic floor therapists in the greater Milwaukee Wisconsin region through a "Pelvic Floor Study Group" list informing them of the need for subjects with this diagnosis so that they may inform their clients of the availability of such research. These clients may then request a referral from their private health care provider.

The pilot study will be completed in twelve months following the commitment of ProHealth Care, Inc. Institutional Review Board as well as procurement of initial funding through grants applied for during 2013. There will be 10 patients enrolled in the pilot study.

Patients will be screened after they are referred by their physician for physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* • Female

  * 18 years or older
  * Current diagnosis of provoked or non-provoked vulvar vestibulitis made by a suitably qualified medical professional
  * Vulvar pain is chronic, defined as having been present for at least 3 months.
  * Visual Analog Score for typical vulvar pain is at least 30/100 Patient has been stabilized on all hormonal interventions (i.e., birth control pills, topical or oral estrogen agents) and will not be altered for the course of the treatment protocol of this study.
  * Subject is willing and able to decrease use of current pain relief medication to manage vulvar pain throughout study participation, and is willing and able to refrain from engaging in other non-study treatments to manage her vulvar vestibulitis symptoms

Exclusion Criteria:

* • Vulvar dermatoses such as lichen sclerosis, squamous cell hyperplasia, or lichen planus

  * Active vaginal or pelvic infection, herpetic infections, vulvar cancer and/or treatment for cancer
  * Previous vestibulectomy or other surgical or procedural interventions (for vestibulitis ) to the treatment area
  * Active infection, wound or other external trauma to the areas to be treated with the laser
  * Other neurological disorders such as Multiple Sclerosis
  * Photosensitivity disorder
  * Pregnant or planning pregnancy prior to study end
  * Serious mental health illness, developmental disability or cognitive impairment that may preclude adequate comprehension of the consent form or ability to record study measures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda A LaBorde, BS PT, Principal Investigator — ProHealth Care, Inc

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cold Laser Treatment: Cold laser used off of the body over the vulvar involved area. The device to be used in this study is the Erchonia Corporation variable frequency pulsed wave low level laser device employing three independent 7 mW, 635 nm red light diodes mounted in a hand-held device and is a variable frequency pulsed wave device. Weekly visits x 6 with 5 minute treatments over vulva and sacral nerve roots each.
  Cold laser: Erchonia Corporation variable frequency pulsed wave low level laser device employing three independent 7 mW, 635 nm red light diodes mounted in a hand-held device and is a variable frequency pulsed wave device.
Period: Overall Study
Arm/Group | Cold Laser Treatment
Started | 10
Completed | 7 (3 did not complete study.)
Not Completed | 3
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: seven completed study and three withdrew
Groups:
- Cold Laser Recipients: 10 enrolled in the study. Seven completed the study and three withdrew. Each participant received six cold laser light therapy treatments and were assessed pre and post treatment with Q tip testing at each treatment visit. There was also a two week follow up scheduled for re-assessment.
  Treatment for each patient was not standardized since there were four therapists involved in data collection and treatment. The treatments included manual therapy mobilizations, neuromuscular rehabilitation with or without EMG biofeedback, home care training which may have included lubricant usage, dilator training, and exercises for the pelvic floor as well as methods of pain relieving modalities.
Arm/Group | Cold Laser Recipients
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Improvement Change in Visual Analogue Pain Scale (VAS) Calculated With Q-tip Palpation Over 6 Sites From Baseline Visit to Follow up at Two Week From Last Visit
Description: III. Q-tip testing:
  . Q-tip pressure will be applied at the following areas, in the exact order listed: 2:00, 10:00, 5:00, 7:00, 12:00, and 6:00. An average VAS report of pain taken overall and compared from first baseline visit to end of study re-assessment two weeks following last treatment.
  • Pain intensity marked an a line with a point between 0-100 on the Visual Analogue Scale (VAS). A separate rating is recorded for each of the 6 numbered areas (see box 1 for reference). 100 is maximum pain level and 0 is no pain measured in centimeters per FDA guidelines for pain calculation on the VAS
Time Frame: Average of all sites Compared from baseline visit and at 8 week (from start) follow up
Measure: Mean (Standard Deviation); unit: percent change from first to last Rx
Arm/Group | Cold Laser Treatment
Number analyzed (Participants) | 7
percent change from first to last Rx | 76.52 (24.36)

2. Secondary Outcome: Change in Patient Specific Functional Scale Questionnaire
Description: Questionnaire that measures on a 0-10 scale (0= No function, and 10= normal function) one function that most impacts the patient's present symptoms (vaginal penetration/intercourse chosen as most important and pertinent) Measured amount of point change on the scale.
Time Frame: Baseline, and two weeks following last treatment at Week 8
Population: women average 26+/- 5.533 Years of age who were not pregnant with appropriate diagnoses
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cold Laser Treatment
Number analyzed (Participants) | 7
units on a scale | 5.25 (1.15)

3. Other Pre Specified Outcome: Change in the Vulvar Pain Functional Scale Questionnaire
Description: Questionnaire of eleven questions involving specific functions that may impart pain in the vulvar region and patient response to present tolerance level. Questions have 4-5 answer choices weighted on a 0-3 scale of impairment, with 3 being worst.
  Worst reported score of functional impact =33. No functional impact = 0
Time Frame: Baseline, and after last treatment visit at Week 8
Population: women average age of 26 +/- 5.533 Years with appropriate diagnoses
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Cold Laser Recipients: 10 enrolled in the study. Seven completed the study and three withdrew. Each participant received six cold laser light therapy treatments and were assessed pre and post treatment with Q tip testing. There was a two week follow up scheduled for assessment.
  Treatment for each patient was not standardized since there were four therapists involved in data collection and treatment. The treatments included manual therapy mobilizations, neuromuscular rehabilitation with or without EMG biofeedback, home care training which may have included lubricant usage, dilator training, and exercises for the pelvic floor as well as methods of pain relieving modalities.
Arm/Group | Cold Laser Recipients
Number analyzed (Participants) | 7
percent change | 32.89 (2.63)

ADVERSE EVENTS:
Groups:
- Cold Laser Light Therapy: The laser unit emits three independent 7 mW, 635 nm red light diodes in a hand-held device and is a variable frequency pulsed wave device. Erchonia low level lasers have been determined safe and effective and non-significant risk (NSR) by the Food and Drug Administration (FDA) for application for numerous and various pain reduction indications, providing justification for the anticipated safety and effectiveness of application The cold laser was administered over 10 minutes as follows: 5 minutes at the area of sacral nerve roots 2-4 in the side-lying position- hertz settings: 14, 8, 12, 28; and 5 minutes at the vulva in the lithotomy position, hertz settings 2: 9,16,33,60 while the outer labia were held open by the therapist. A sweeping motion was used during administration. The laser head was positioned approximately 3 inches from the skin surface and did not touch the skin. The patient wore safety goggles while the laser treatment was provided.
Arm/Group | Cold Laser Light Therapy
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed were the choice of the participant to end participation. One participant became pregnant during the study. Other reasons were related to participant cost of healthcare visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No